CLINICAL TRIAL: NCT01907269
Title: Activating Patients to Reduce OsteoPOrosiS
Brief Title: A Direct-to-patient Intervention to Increase Rates of Osteoporosis Care
Acronym: APROPOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Massachusetts, Worcester (Other); Helen Hayes Hospital (Other); Kaiser Permanente (Other); Cedars-Sinai Medical Center (Other); University of Pittsburgh (Other); University of Cincinnati (Other)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: X110928001; R01AR060240 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Video-based intervention (Experimental): Video-based intervention providing personalized feedback regarding patients' risk of subsequent fractures, customized information regarding osteoporosis care, and messaging to activate patients to become more engaged in improving osteoporosis treatment and doctor-patient communication. This novel content will use "story-telling" delivered via the Internet and DVDs. The content will be uniquely tailored to each person based on their reported barriers to care, age and race/ethnicity. The video-based intervention materials will be augmented by a personal phone call and interactive voice response messaging.
  Interventions: Behavioral: Video-based Intervention
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Video-based Intervention — Video clips delivered by DVD and Internet
  Arms: Video-based intervention

SUMMARY:
The purpose of this study is to conduct a randomized trial of a tailored intervention designed to provide personalized feedback regarding patients' risk of subsequent fractures, customized information regarding osteoporosis care, and messaging to activate patients to become more engaged in improving osteoporosis treatment and doctor-patient communication. This novel content will use "story-telling" delivered via the Internet and digital video discs (DVDs). The content will be uniquely tailored to each person based on barriers to care, age and race/ethnicity. We will conduct a controlled, cluster-randomized trial of this intervention to determine differences in post-intervention rates of osteoporosis care between two randomization arms.

We hypothesize that participants randomized to the intervention arm, compared to those randomized to a control arm, will receive more osteoporosis care at 6 months post-intervention, as evidenced by higher rates of: (H1) Prescription osteoporosis therapies, (H2) Non-prescription therapy with calcium and vitamin D, and (H3) Bone mineral density (BMD) testing.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of fracture

Exclusion Criteria:

* Self-reported current prescription osteoporosis treatment

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2684 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Saag, MD, MSc, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Massachusetts at Worcester, Worcester, Massachusetts
  - New York University, New York, New York
  - Jewish Hospital of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Group Health Research Institute, Seattle, Washington

REFERENCES:
- [Background] Yood RA, Mazor KM, Andrade SE, Emani S, Chan W, Kahler KH. Patient decision to initiate therapy for osteoporosis: the influence of knowledge and beliefs. J Gen Intern Med. 2008 Nov;23(11):1815-21. doi: 10.1007/s11606-008-0772-0. Epub 2008 Sep 12. PMID 18787907
- [Background] Weinstein ND. The precaution adoption process. Health Psychol. 1988;7(4):355-86. doi: 10.1037//0278-6133.7.4.355. PMID 3049068
- [Result] Danila MI, Outman RC, Rahn EJ, Mudano AS, Thomas TF, Redden DT, Allison JJ, Anderson FA, Anderson JP, Cram PM, Curtis JR, Fraenkel L, Greenspan SL, LaCroix AZ, Majumdar SR, Miller MJ, Nieves JW, Safford MM, Silverman SL, Siris ES, Solomon DH, Warriner AH, Watts NB, Yood RA, Saag KG. A multi-modal intervention for Activating Patients at Risk for Osteoporosis (APROPOS): Rationale, design, and uptake of online study intervention material. Contemp Clin Trials Commun. 2016 Dec 15;4:14-24. doi: 10.1016/j.conctc.2016.06.010. PMID 27453960
- [Result] Danila MI, Outman RC, Rahn EJ, Mudano AS, Redden DT, Li P, Allison JJ, Anderson FA, Wyman A, Greenspan SL, LaCroix AZ, Nieves JW, Silverman SL, Siris ES, Watts NB, Miller MJ, Curtis JR, Warriner AH, Wright NC, Saag KG. Evaluation of a Multimodal, Direct-to-Patient Educational Intervention Targeting Barriers to Osteoporosis Care: A Randomized Clinical Trial. J Bone Miner Res. 2018 May;33(5):763-772. doi: 10.1002/jbmr.3395. Epub 2018 Feb 26. PMID 29377378

RESULTS

PARTICIPANT FLOW:
Period: 6 Month Outcome Measures Post-interventi
Arm/Group | Video-based Intervention | Usual Care
Started | 1342 | 1342
Completed | 953 | 1053
Not Completed | 389 | 289
Period: 18 Month Outcome Measures Post-intervent
Arm/Group | Video-based Intervention | Usual Care
Started | 1178 | 1250
Completed | 859 | 970
Not Completed | 319 | 280

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video-based Intervention | Usual Care | Total
Number analyzed (Participants) | 1342 | 1342 | 2684
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (8) | 74.9 (7.9) | 74.9 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1342 | 1342 | 2684
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 21 | 46
  Not Hispanic or Latino | 1317 | 1321 | 2638
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 13 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 52 | 98
  White | 1247 | 1239 | 2486
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 36 | 38 | 74
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1342 | 1342 | 2684
Number of Participants who Completed Barriers to Osteoporosis Treatment [Count of Participants; unit: Participants] — A list of seven potentially modifiable barriers was presented to patients in the baseline survey. Those that ranked them in the intervention arm (N=482) were allocated a tailored online and video intervention based on their response. Unfortunately, not all participants ranked barriers (i.e., they didn't follow the survey directions). Individuals that did not rank barriers received an intervention corresponding to the next level of tailoring (e.g., Responses on the Patient's Views about Osteoporosis Use and Therapy Scale, Readiness to Behavior Change, or Osteoporosis treatment history). Population: Data were only evaluated for intervention tailoring on the "Video-based intervention" arm. "Usual care" data on this measure was not evaluated for the purposes of tailoring, therefore the Row population consists only of the intervention arm (n=1342) and does not include usual care. This results in the row population differing from overall.
  Participants
    number analyzed (Participants) | 1342 | 0 | 1342
    (all) | 482 | 0 | 482
Number of Participants who completed Patient's Views about Osteoporosis and Use of Therapy Scale [Count of Participants; unit: Participants] — Patients in the "Video-based intervention" arm that didn't rank barriers, but who did complete the Patient's Views about Osteoporosis and Use of Therapy Scale (N=429) received a tailored intervention based on responses to this scale. Unfortunately, not all participants completed the Patient's Views about Osteoporosis and Use of Therapy Scale (i.e., they didn't follow the survey directions); these individuals received an intervention corresponding to the next level of tailoring (e.g., Readiness to Behavior Change, or Osteoporosis treatment history). Population: Data were only evaluated for intervention tailoring on the "Video-based intervention" arm. "Usual care" data on this measure was not evaluated for the purposes of tailoring, therefore the Row population consists only of the intervention arm (n=1342) and does not include usual care. This results in the row population differing from overall.
  Participants
    number analyzed (Participants) | 1342 | 0 | 1342
    (all) | 429 | 0 | 429
Number of Participants who Completed Readiness to Behavior Change [Count of Participants; unit: Participants] — Patients in the "Video-based intervention" arm that didn't rank barriers,and did not complete the Patient's Views about Osteoporosis and Use of Therapy Scale received a tailored intervention based on their readiness to behavior change (N=300) as assessed by a modified version of Weinstein's Precaution Adoption Process Model. Unfortunately, not all participants completed the Readiness to Behavior Change (i.e., they didn't follow the survey directions); these individuals received an intervention corresponding to the next level of tailoring (e.g., Osteoporosis treatment history). Population: Data were only evaluated for intervention tailoring on the "Video-based intervention" arm. "Usual care" data on this measure was not evaluated for the purposes of tailoring, therefore the Row population consists only of the intervention arm (n=1342) and does not include usual care. This results in the row population differing from overall.
  Participants
    number analyzed (Participants) | 1342 | 0 | 1342
    (all) | 300 | 0 | 300
Number of Participants who Completed the Osteoporosis Treatment History (tailoring) [Count of Participants; unit: Participants] — Patients in the "Video-based intervention" arm that didn't rank barriers, did not complete the Patient's Views about Osteoporosis and Use of Therapy Scale, and where readiness to behavior change could not be assessed received an intervention tailored based on their osteoporosis treatment history as assessed by our survey (N=131). The categorization for this variable was dichotomous, those that indicated they had received previous treatment or those that indicated they had not received previous treatment. Population: Data were only evaluated for intervention tailoring on the "Video-based intervention" arm. "Usual care" data on this measure was not evaluated for the purposes of tailoring, therefore the Row population consists only of the intervention arm (n=1342) and does not include usual care. This results in the row population differing from overall.
  Participants
    number analyzed (Participants) | 1342 | 0 | 1342
    (all) | 131 | 0 | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Initiate an Osteoporosis Prescription Medication
Description: We will assess the number of participants that self-report the initiation of an osteoporosis prescription medication. It will be assessed using a self-completed survey. Osteoporosis prescription medications that will be assessed include: alendronate, calcitonin, denosumab ibandronate, raloxifene, risedronate, teriparatide, and zoledronic acid. We will not include initiation of estrogen hormone therapies as part of the primary outcome.
Time Frame: 6 months post-intervention
Population: For the Intent-to-Treat Analysis the data was imputed for non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based Intervention | Usual Care
Number analyzed (Participants) | 1342 | 1342
Participants | 157 | 153

2. Secondary Outcome: Number of Participants Who Reported Use of Calcium and Vitamin D
Description: We will assess the use of calcium and vitamin D by participant. This will be assessed on a self-completed survey. Participants will be asked if they are currently taking a calcium supplement and/or vitamin D supplement.
Time Frame: 6 and 18 months post-intervention
Population: For the Intent-to-Treat Analysis the data was imputed for non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based Intervention | Usual Care
Number analyzed (Participants) | 1342 | 1342
Participants
  Vitamin D (6 months) | 554 | 562
  Calcium (6 months) | 427 | 437
  Vitamin D (18 months): number analyzed (Participants) | 1178 | 1250
  Vitamin D (18 months) | 475 | 572
  Calcium (18 months): number analyzed (Participants) | 1178 | 1250
  Calcium (18 months) | 249 | 310

3. Secondary Outcome: Number of Participants Who Reported Receipt of Bone Mineral Density (BMD) Testing
Description: Self-report of a receipt of a DXA scan (Bone Mineral Density test).
Time Frame: 6 and 18 months post-intervention
Population: For the Intent-to-Treat Analysis the data was imputed for non-responders. Surveys for BMD (18 months) included 3 responses. If participants marked option (2) that they had received a BMD, but > 12 months ago they were excluded from analyses. Thus our overall population analyzed (those marking response 1 or 3) is different than our participant flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based Intervention | Usual Care
Number analyzed (Participants) | 1342 | 1342
Participants
  BMD (6 months): number analyzed (Participants) | 469 | 469
  BMD (6 months) | 290 | 268
  BMD (18 months): number analyzed (Participants) | 643 | 663
  BMD (18 months) | 530 | 522

4. Secondary Outcome: Number of Participants That Initiate an Osteoporosis Prescription Medication
Description: We will assess the number of participants that self-report the initiation of an osteoporosis prescription medication. It will be assessed using a self-completed survey. Osteoporosis prescription medications that will be assessed include: alendronate, calcitonin, denosumab ibandronate, raloxifene, risedronate, teriparatide, and zoledronic acid. We will not include initiation of estrogen hormone therapies as part of the outcome.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based Intervention | Usual Care
Number analyzed (Participants) | 1178 | 1250
Participants | 136 | 131

5. Other Pre Specified Outcome: Number of Participants Who Reported Communicating With a Health Care Provider About Osteoporosis Care
Time Frame: 6 and 18 months post-intervention
Population: For the Intent-to-Treat Analysis the data was imputed for non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based Intervention | Usual Care
Number analyzed (Participants) | 1342 | 1342
Participants
  Bone health discussion w/provider (6 months) | 583 | 573
  Bone health discussion w/provider (18 months): number analyzed (Participants) | 1178 | 1250
  Bone health discussion w/provider (18 months) | 779 | 806

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Video-based Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Low rates of osteoporosis treatment initiation; Self-reported fracture history subject to recall bias; Low % of participants reported fracture in 12-months prior to intervention; Low % of participants who interacted with intervention appreciably

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No